CLINICAL TRIAL: NCT05984771
Title: Efficacy and Safety of the Combination of Superoxide Dismutase, Alpha Lipoic Acid, Vitamins B12, B1, B2, B6, E, Mg, Zn and Palmitoylethanolamide for 6 Months in Patients With Diabetic Neuropathy : A Pilot Study
Brief Title: Efficacy and Safety of the Combination of Ten Elements for 6 Months in Patients With Diabetic Neuropathy : A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Prof. Triantafyllos Didangelos, Professor of Internal Medicine and Diabetology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 54230/12.12.2020
Record Dates: First submitted 2023-06-26; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Neuropathies; Diabetes Mellitus; Dietary Supplement
Keywords: diabetes mellitus; neuropathy; pain
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain

STUDY DESIGN:
Intervention Model Description: pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator and examiner did not know the type of drug provided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): 10-element combination tablet (n=30) Superoxide Dismutase (SOD, 70 UI), Palmitoylethanolamide (PEA, 300 mg) Alpha Lipoic Acid (ALA, 300 mg), vitamins B6 (1.5 mg), B1 (1.1 mg), B12 (2.5 mcg), E (7.5 mg), Nicotinamide (9 mg) and minerals (Mg 30 mg, Zn 2,5 mg) in one tablet for 6 months
  Interventions: Dietary Supplement: Epineuron
- Placebo (Placebo Comparator): usual care
  Interventions: Other: Placebo group

INTERVENTIONS:
Dietary Supplement: Epineuron — Superoxide Dismutase (SOD, 70 UI), Palmitoylethanolamide (PEA, 300 mg) Alpha Lipoic Acid (ALA, 300 mg), vitamins B6 (1.5 mg), B1 (1.1 mg), B12 (2.5 mcg), E (7.5 mg), Nicotinamide (9 mg) and minerals (Mg 30 mg, Zn 2,5 mg) in one tablet (Epineuron)
  Arms: Active group
Other: Placebo group — Usual care
  Arms: Placebo

SUMMARY:
To investigate the efficacy of Superoxide Dismutase (SOD, 70 UI), Palmitoylethanolamide (PEA, 300 mg) Alpha Lipoic Acid (ALA, 300 mg), vitamins B6 (1.5 mg), B1 (1.1 mg), B12 (2.5 mcg), E (7.5 mg), Nicotinamide (9 mg) and minerals (Mg 30 mg, Zn 2,5 mg) in one tablet in patients with Diabetic Neuropathy (DN).

DETAILED DESCRIPTION:
To investigate the efficacy of Superoxide Dismutase (SOD, 70 UI), Palmitoylethanolamide (PEA, 300 mg) Alpha Lipoic Acid (ALA, 300 mg), vitamins B6 (1.5 mg), B1 (1.1 mg), B12 (2.5 mcg), E (7.5 mg), Nicotinamide (9 mg) and minerals (Mg 30 mg, Zn 2,5 mg) in one tablet in patients with Diabetic Neuropathy (DN).

Patients - methods: In this pilot study, 61 patients with Diabetes Mellitus Type 2 (DMT2, 31 women), with mean duration of DM 17.5 years and mean age 63 years were randomly assigned, either to receive the combination of ten elements (2 tablets/24h) in the active group, (n=30), or the placebo (n=31) for 6 months. We used Michigan Neuropathy Screening Instrument Questionnaire and Examination (MNSIQ and MNSIE), measured vibration perception threshold (VPT) and Cardiovascular Autonomic Reflex Tests (CARTs). Nerve function was assessed by DPN Check [sural nerve conduction velocity (SNCV) and amplitude (SNAP)]. Sudomotor function was assessed with SUDOSCAN that measures electrochemical skin conductance in hands and feet (ESCH and ESCF). Pain (PS) questionnaire was administered, also. All patients received metformin for at least 4 years.

ELIGIBILITY:
Inclusion Criteria:

* on metformin therapy for at least 4 years
* diabetes mellitus type 2 with diabetic neuropathy
* painful neuropathy

Exclusion Criteria:

* healthy
* without diabetic neuropathy
* pregant

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Nerve conduction study to measure the velocity of the nerve impulse in the sural nerve | 6 months
  Measurement of nerve conduction velocity with Neurometrix Diabetic Peripheral Neuropathy scan device
Measurement of individual Vibration Perception Threshold to study vibration perception in the feet | 6 months
  Measurement of vibration perception threshold with Biothesiometer
Michigan Screening Neuropathy Questionnaire and Examination | 6 months
  use of michigan screening questionnaire and examination
Measurement of electrochemical skin conductance | 6 months
  measurement with Sudoscan the electrochemical skin conductance in hands and feet

SECONDARY OUTCOMES:
Glycated Hemoglobin | 6 months
  Measurement of Glycated Hemoglobin
vitamin B12 levels | 6 months
  measurement of B12 levels

CONTACTS AND LOCATIONS:
Locations (1):
- University General Hospital AHEPA, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No